CLINICAL TRIAL: NCT00065221
Title: Trial of Encapsulated Ginger as a Treatment for Chemotherapy-Induced Nausea and Vomiting
Brief Title: Ginger Control of Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001735-01 (NIH)
Record Dates: First submitted 2003-07-18; First posted 2003-07-22 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Nausea; Vomiting; Chemotherapy
Keywords: Ginger; Plant preparation; Herbal medicine; Chemotherapy; Nausea
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

INTERVENTIONS:
Drug: Ginger

SUMMARY:
This is a trial to determine the safety and efficacy of ginger in reducing the prevalence and severity of chemotherapy induced nausea and vomiting.

DETAILED DESCRIPTION:
Chemotherapy induced nausea and vomiting significantly reduces patients' quality of life, increases fatigue, anxiety, and increases costs of health care delivery. Ginger (Zingiber officinalis) is already used in traditional folk medicine to treat nausea and vomiting in various populations. Ginger's ability to block 5-HT3 receptors and its free-radical scavenging in the intestines suggest that it may be beneficial for reducing both the prevalence and severity of chemotherapy induced nausea and vomiting. Despite ginger's possible benefits in reducing the prevalence and severity of chemotherapy induced nausea and vomiting, no dosing and/or safety studies have been performed.

This study will assess the efficacy and safety of two dose levels (1000 mg, or 2000 mg, orally/day) of Zingiber officinalis extract (standardized for 5% gingerols) in patients undergoing chemotherapy (cisplastin or adriamycin) who have experienced at least one episode of chemotherapy induced nausea and vomiting despite optimal conventional medical therapy. The primary aim of the study is to determine the most efficacious dose of powdered ginger-root for reducing the prevalence and severity of acute nausea and vomiting. Secondary aims of the study include (1) determination of the most efficacious dose of powdered ginger-root for reducing the prevalence and severity of delayed nausea and vomiting; (2) assessment of the safety of different doses of oral powdered ginger root in patients receiving chemotherapy; and (3) determination if study participants can discern if they are receiving placebo or ginger. Participants receiving either adriamycin or cisplatin for cancer related treatment will be randomized to receive one of two doses of powdered ginger or placebo immediately prior to chemotherapy infusion. Participants will be followed for 72 hours after infusion in order to assess frequency and severity of nausea and vomiting. Baseline and 72 hour post chemotherapy labs will be used to assess safety profile of ginger.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of cancer and currently receiving chemotherapy
* Currently being treated with any chemotherapeutic agent at any dose, and have experienced nausea and/or vomiting from a previous round of chemothearpy
* Scheduled to receive a 5-HT3 receptor antagonist antiemetic: ondansetron (Zofran®) granistron (Kytril®), tropisetron (Navoban®) or dolasetron mesylate (Anzemet®), palanosetron (Alozi) and/or the NK1 antagonist aprepitant (Emend)
* Must be able to swallow capsules
* Must be able to understand English or Spanish, complete questionnaires in English or Spanish
* Women of childbearing age to use appropriate birth control

Exclusion criteria:

* Chemotherapy regimens with multiple-day doses
* Clinical evidence of current or impending bowel obstruction or symptomatic brain metastases

  * Concurrent radiotherapy that is classified as high or intermediate risk of causing nausea and vomiting; total body irradiation, hemi-body, upper abdomen, abdominal-pelvic mantle, cranium, craniospinal irradiation
* Pregnant or lactating
* Patients with a history of a bleeding disorder(s) or those experiencing thrombocytopenia
* Currently be taking ginger or have taken ginger in the last month
* Have an allergy to ginger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (6):
- United States (5):
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - University of Michigan Cancer Center Complementary and Alternative Medicine Research Center, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Community Clinic Oncology Program, Grand Rapids, Michigan
  - Our Lady of Mercy Medical Center, Comprehensive Cancer Center, The Bronx, New York
- Community Clinic Oncology Program, San Juan, Puerto Rico